CLINICAL TRIAL: NCT00396201
Title: Treatment With AMD3100 Added to a Mobilizing Regimen of G-CSF to Increase the Number of Peripheral Blood Stem Cells in Patients With Hodgkin's Disease
Brief Title: AMD3100 (Plerixafor) Added to a Mobilizing Regimen of Granulocyte-colony Stimulating Factor (G-CSF) to Increase the Number of Peripheral Blood Stem Cells (PBSCs) in Patients With Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2106
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin's Disease; Stem cell mobilization; apheresis
MeSH Terms: conditions — Hodgkin Disease | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants with Hodgkin's Disease (HD) (Experimental): Participants with Hodgkin's Disease who were eligible for autologous peripheral blood stem cell transplantation.
  Interventions: Drug: G-CSF Plus Plerixafor

INTERVENTIONS:
Drug: G-CSF Plus Plerixafor — Randomized participants underwent mobilization with G-CSF 10 µg/kg/day for 4 days, administered by subcutaneous injection (SC) injection. On the evening of Day 4, participants received a dose of plerixafor 240 µg/kg, administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF 10 µg/kg and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor (within 60 minutes after administration of G-CSF). Participants continued to receive an evening dose of plerixafor followed the next day by a morning dose of G-CSF and apheresis for up to a maximum of 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Other Names: Mozobil; AMD3100

SUMMARY:
Participants with Hodgkin's Disease (HD) who have been treated with cyto-reductive chemotherapy, who are to undergo autologous stem cell transplantation, and who meet the inclusion/exclusion criteria are eligible to enter this efficacy, safety and pharmacokinetic (PK) study. The only changes to the standard of care is the addition of plerixafor to a granulocyte-colony stimulating factor (G-CSF) mobilization regimen on each day prior to apheresis. The purpose of this protocol is to determine the proportion of participants who reach a target number of CD34+ stem cells (≥5*10^6 cells/kg) after hematopoietic stem cell mobilization with G-CSF and plerixafor. Safety and PK parameters are also collected.

DETAILED DESCRIPTION:
Participants with HD who have been treated with cyto-reductive chemotherapy, who are to undergo autologous stem cell transplantation, and who meet the inclusion/exclusion criteria are eligible to enter this study. The only changes to the standard of care is the addition of plerixafor to a G-CSF mobilization regimen on the day prior to apheresis and the collection of blood samples for pharmacokinetic (PK) analysis and pharmacodynamics (PD) analysis by CD34+ fluorescence-activated cell sorting (FACS) analysis. Blood samples for PK and CD34+ FACS analyses will be obtained prior to and after the first dose of plerixafor. Participants will undergo mobilization with G-CSF (10 µg/kg daily) and will receive plerixafor (240 µg/kg) on each day prior to apheresis. Participants will be apheresed for up to 5 consecutive days in order to collect the target number of CD34+ stem cells, (≥5*10^6 cells/kg). After apheresis, all participants will be treated with high dose chemotherapy in preparation for transplantation. Participants will be transplanted with cells obtained from the G-CSF plus plerixafor mobilization regimen. In the event that a sufficient number of cells for transplantation are not obtained from the collection, cells may be retained and pooled for transplantation at the investigator's discretion.

The primary endpoint is the proportion of HD participants who collect ≥5*10^6 CD34+ cells/kg with this mobilization regimen. The secondary endpoints include the safety of this mobilization regimen, the proportion of participants who collect ≥2*10^6 CD34+ cells/kg, the change in CD34+ cells circulating in the peripheral blood after a dose of plerixafor, and the number of days of apheresis required to obtain ≥5*10^6 CD34+ cells/kg. In addition, success of the transplantation will be evaluated by measuring the time to engraftment of PMNs and PLTs. Participants will be followed for 12 months to assess transplant durability.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD eligible for autologous transplantation
* No more than 3 prior regimens of chemotherapy (Rituximab is not considered chemotherapy for the purpose of this study.)
* 4 weeks since last cycle of chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* The patient has recovered from all acute toxic effects of prior chemotherapy
* White blood cell count (WBC) >3.0*10^9/L
* Absolute polymorphonuclear cells (PMN) count >1.5*10^9/L
* Platelet (PLT) count >100*10^9/L
* Serum creatinine ≤2.2 mg/DL
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 x upper limit of normal (ULN)
* Left ventricle ejection fraction >45% by normal echocardiogram or multiple-gated acquisition (MUGA) scan
* Forced expiratory volume of the lung in the first second (FEV1) >60% of predicted or diffusing capacity of the lung for carbon monoxide (DLCO) >45% of predicted
* Negative for human immunodeficiency virus (HIV)

Exclusion Criteria:

* A co-morbid condition which, in the view of the investigator, renders the patient at high risk for treatment complications
* Patients who have failed previous collections
* A residual acute medical condition resulting from prior chemotherapy
* Hodgkin's disease involving the central nervous system
* Acute infection
* Fever (temp >38°C/100.4°F)
* Patients whose actual body weight exceeds 150% of their ideal body weight
* History of ventricular arrhythmias
* History of paresthesias
* Patients who previously received experimental therapy within 4 weeks of enrolling in this study or who are currently enrolled in another experimental study during the mobilization period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-11; Primary Completion 2006-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Washington University School of Medicine,Division of Bone Marrow Transplantation & Leukemia, St Louis, Missouri, United States

REFERENCES:
- [Background] Cashen A, Lopez S, Gao F, Calandra G, MacFarland R, Badel K, DiPersio J. A phase II study of plerixafor (AMD3100) plus G-CSF for autologous hematopoietic progenitor cell mobilization in patients with Hodgkin lymphoma. Biol Blood Marrow Transplant. 2008 Nov;14(11):1253-61. doi: 10.1016/j.bbmt.2008.08.011. PMID 18940680

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hodgkin's Disease (HD): Participants with Hodgkin's disease who were eligible for autologous peripheral blood stem cell transplantation. Participants underwent mobilization with granulocyte-colony stimulating factor (G-CSF) [10 µg/kg each day (QD)] and received plerixafor (240 µg/kg) on each day prior to apheresis. Participants were apheresed for up to 5 consecutive days in order to collect the target number of CD34+ stem cells, (≥5*10^6 cells/kg).
Period: Treatment Period
Arm/Group | Participants With Hodgkin's Disease (HD)
Started | 22
Completed | 22 (Completed refers to completed all treatment visits.)
Not Completed | 0
Period: Follow-up Period
Arm/Group | Participants With Hodgkin's Disease (HD)
Started | 21 (Participants who had transplants. One had insufficient collection of cells so no transplant.)
Completed | 21 (Follow-up visit 12 months post-transplant)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Hodgkin's Disease (HD): Participants with Hodgkin's Disease who were eligible for autologous peripheral blood stem cell transplantation. Participants underwent mobilization with G-CSF (10 µg/kg QD) and received plerixafor (240 µg/kg) on each day prior to apheresis. Participants were apheresed for up to 5 consecutive days in order to collect the target number of CD34+ stem cells, (≥5*10^6 cells/kg).
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 22

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieved ≥5*10^6 CD34+ Cells/kg Following Treatment With Plerixafor and G-CSF
Description: The proportion of total participants who mobilized ≥5*10^6 CD34+ cells/kg based on data from local laboratories.
Time Frame: Day 5 up to Day 9
Population: Intent to treat population which included all participants who received plerixafor.
Measure: Number; unit: proportion of participants
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 22
proportion of participants
  Proportion achieving ≥5*10^6 CD34+ cells/kg | 0.68
  Proportion not achieving ≥5*10^6 CD34+ cells/kg | 0.32

2. Secondary Outcome: Overall Participant Counts of Adverse Events During the Treatment Period
Description: Adverse Events were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe and life-threatening) and relatedness (5 steps from 'not related' to 'definitely related') to study treatment. Time frame starts on the first day of G-CSF mobilization to the day prior to chemotherapy/ablative treatment in preparation for transplant.
  See the separate Serious Adverse Event section for a summary of AEs the investigator assessed as serious.
Time Frame: Day 0 - approximately day 38
Population: Safety population consisting of all participants who received G-CSF and/or plerixafor.
Measure: Number; unit: participants
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 22
participants
  Reporting at least one AE | 17
  Severity - Mild | 5
  Severity - Moderate | 11
  Severity - Severe | 1
  Severity - Life Threatening | 0
  Relationship - Not Related | 2
  Relationship - Probably Not Related | 1
  Relationship - Possibly Related | 12
  Relationship - Probably Related | 1
  Relationship - Definitely Related | 1

3. Secondary Outcome: Proportion of Participants Who Achieved ≥2*10^6 CD34+ Cells/kg Following Treatment With Plerixafor and G-CSF
Description: The proportion of total participants who mobilized ≥2*10^6 CD34+ cells/kg based on data from local laboratories.
Time Frame: Day 5 up to day 9
Population: Intent to treat population which included all participants who received plerixafor.
Measure: Number; unit: proportion of participants
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 22
proportion of participants
  Proportion achieving ≥2*10^6 CD34+ cells/kg | 0.95
  Proportion not achieving ≥2*10^6 CD34+ cells/kg | 0.05

4. Secondary Outcome: Fold (Relative) Increase in Peripheral Blood (PB) CD34+ Cells/µL
Description: The fold increase was measured by fluorescence activated cell sorting (FACS) analysis using local laboratory data and was expressed as a ratio. Fold increase = (pre-apheresis PB CD34+ cells/µL)/(pre-plerixafor dosing PB CD34+ cells/µL).
Time Frame: Days 4-5 (first dose of plerixafor to apheresis)
Population: Intent to treat population which included all participants who received plerixafor and had pre- and post-plerixafor CD34+ cell counts available; 3 participants had missing results data and were not included.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 19
ratio | 3.2 (1.1)

5. Secondary Outcome: Participant Counts Grouped by Number of Apheresis Days Required to Collect ≥ 5*10^6 CD34+ Cells/kg
Description: Counts of participants grouped by the number of apheresis days needed to collect a target for transplantation of ≥5*10^6 CD34+ cells/kg as determined by local laboratory data.
Time Frame: Day 5 up to day 9
Population: Intent to treat population which included all participants who received plerixafor and achieved a target of ≥5*10^6 CD34+cells/kg
Measure: Number; unit: participants
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 15
participants
  1 day of apheresis | 7 (0.9) [1.0 to 3.0]
  2 days of apheresis | 6
  3 days of apheresis | 2

6. Secondary Outcome: Number of Days Post-Transplantation to Polymorphonuclear Leukocyte (PMN) Engraftment
Description: Median number of days to PMN engraftment following transplantation. Engraftment was defined as PMN counts ≥ 0.5*10^9/L for 3 consecutive days or ≥ 1.0*10^9/L for 1 day. Time to engraftment corresponded to the first day that the criteria were met.
Time Frame: Up to Month 13 (up to 12 months post transplant)
Population: Intent to treat population which included all participants who received plerixafor and had a transplant.
Measure: Median (Full Range); unit: days
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 21
days | 9.0 (1.2) [8.0 to 14.0]

7. Secondary Outcome: Number of Days Post Transplantation to Platelet (PLT) Engraftment
Description: Median number of days to PLT engraftment following transplantation. Engraftment success was evaluated according to local site practice. Time to engraftment corresponded to the first day that criteria were met.
Time Frame: Up to Month 13 (up to 12 months post transplant)
Population: Intent to treat population which included all participants who received plerixafor and had a transplant. One participant's time to engraftment was unknown due to missing lab values.
Measure: Median (Full Range); unit: days
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 20
days | 19.0 (3.8) [11.0 to 29.0]

8. Secondary Outcome: Number of Participants With a Durable Graft at 12 Months
Description: Graft durability was assessed by the Investigator based on complete blood count (CBC) and differential analyses at 12 months post transplantation. A graft was considered durable if blood counts were normal (acceptable) and still met the criteria for PLT and PMN engraftment.
Time Frame: 13 months
Population: Intent to treat population which included all participants who received plerixafor and had a transplant.
Measure: Number; unit: participants
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 21
participants | 21

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) Following a Single Dose of Plerixafor
Description: Maximum plasma concentration (Cmax) of plerixafor following the first single dose of 240 ug/kg plerixafor administered.
Time Frame: Day 4
Population: The last nine study participants had pharmacokinetic blood samples taken, as reflected in a protocol amendment. Results include participants from the last nine participants who had the relevant test data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 9
ng/mL | 831 (183)

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) Following a Single Dose of Plerixafor
Description: Time to maximum plasma concentration (Tmax) of plerixafor following the first single dose of 240 ug/kg plerixafor was determined from direct observation of the data.
Time Frame: Day 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 9
hours | 0.6 (0.4)

11. Secondary Outcome: Half-life (T1/2) Following a Single Dose of Plerixafor
Description: Plasma elimination half-life (T1/2) following a single dose of 240 ug/kg plerixafor.
Time Frame: Day 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 8
hours | 3.5 (0.7)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 10 Hours (AUC0-10) Following a Single Dose of Plerixafor
Description: Area under the plasma concentration-time curve from 0 to 10 hours (AUC0-10) following the first single dose of 240 ug/kg plerixafor.
Time Frame: Days 4-5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 9
ng*hr/mL | 3572 (772)

13. Secondary Outcome: Apparent Clearance (CL/F) of Single-dose Plerixafor
Description: Apparent clearance was calculated the mean dose of plerixafor divided by the area under the plasma concentration-time curve from 0 hours to infinity (AUC0-inf).
Time Frame: Day 4-5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 8
mL/hr | 5138 (2029)

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) Following a Single-dose of Plerixafor
Description: The volume of distribution (Vz/F) was calculated as apparent clearance divided by the terminal elimination rate constant.
Time Frame: Day 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Participants With Hodgkin's Disease (HD)
Number analyzed (Participants) | 8
mL | 25464 (9002)

ADVERSE EVENTS:
Time Frame: Day 1 (start of G-CSF Mobilization plus Treatment/Apheresis) to the day before starting chemotherapy. Chemotherapy typically started within 30 days of the last apheresis (which may have occurred on Day 5, 6, 7, or 8).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Each AE table includes all events, regardless of reported relationship to study treatment or grade.
Arm/Group | Participants With Hodgkin's Disease (HD)
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 17/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Hodgkin's Disease (HD) (N=22)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Paraesthesia oral (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Catheter site haematoma (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Catheter site pain (General disorders) | 1
Chills (General disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 5
Feeling hot (General disorders) | 1
Injection site discharge (General disorders) | 1
Injection site erythema (General disorders) | 15
Injection site haemorrhage (General disorders) | 3
Injection site irritation (General disorders) | 1
Injection site swelling (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 5
Nervousness (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pallor (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.